CLINICAL TRIAL: NCT05313490
Title: Exercise Fatiguability in Older Adults: The Protective Effects of Dietary Nitrate Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Timothy Fulton, Principal Investigator, Marquette University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HR-4040
Record Dates: First submitted 2022-02-14; First posted 2022-04-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice (Active Comparator): The subject will ingest 140mL of a nitrate-rich beetroot juice each day for 7 consecutive days.
  Interventions: Dietary Supplement: Beetroot Juice
- Placebo Beetroot Juice (Placebo Comparator): The subject will ingest 140mL of a placebo (nitrate-depleted) beetroot juice each day for 7 consecutive days.
  Interventions: Other: Placebo Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — 7 days of 140 mL per day of beetroot juice
  Other Names: James White Drinks Beet It Sport 400
  Arms: Beetroot Juice
Other: Placebo Beetroot Juice — 7 days of 140 mL per day of placebo beetroot juice
  Arms: Placebo Beetroot Juice

SUMMARY:
Vascular and skeletal muscle function decline with age and are associated with decreased nitric oxide (NO) bioavailability. Dietary nitrate supplementation in the form of beet root juice increases NO bioavailability and improves exercise tolerance in younger adults, yet its effects on fatigability in older adults are largely unknown. The proposed research will investigate the impact of increased NO bioavailability on vascular function, skeletal muscle bioenergetics, and fatigability in older (≥65 yrs) men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥ 60 years old

Exclusion Criteria:

1. body mass index ≥40 kg/m2;
2. type 1 or type 2 diabetes or HbA1c >6.5%
3. uncontrolled hypertension;
4. active cancer, cancer in remission, or having received treatment for any form of cancer in the previous five years;
5. coronary artery disease;
6. cardiovascular disease (e.g., PAD, PVD);
7. abnormal and untreated thyroid function;
8. chronic and/or regular nonsteroidal anti-inflammatory drugs (NSAID) consumption,
9. tobacco use (includes smoking);
10. any condition that presents a limitation to exercise (e.g., severe arthritis, COPD, neuromuscular disorder, moderate or severe cognitive impairment, Alzheimer's Disease, severe untreated sleep apnea).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in fatigability of the knee extensor muscles with beetroot juice supplementation | Day 8 (after 7 days of placebo supplementation) and day 29 (after 14 days of a washout period with no supplementation plus 7 days of beetroot juice supplementation)
  Fatigability will be quantified as the reduction in limb muscle power output during a 4-minute dynamic fatiguing exercise task using a dynamometer. Fatigability after 7 days of beetroot juice supplementation will be compared with fatigability after 7 days of placebo supplementation, with the outcome measure being the change (or difference) between these two supplementation conditions.

SECONDARY OUTCOMES:
Change in femoral artery blood flow with beetroot juice supplementation | Day 8 (after 7 days of placebo supplementation) and day 29 (after 14 days of a washout period with no supplementation plus 7 days of beetroot juice supplementation)
  Femoral artery blood flow will be quantified as the change in femoral artery blood flow during a 4-minute dynamic fatiguing exercise task using a ultrasonography. Femoral artery blood flow after 7 days of beetroot juice supplementation will be compared with Femoral artery blood flow after 7 days of placebo supplementation, with the outcome measure being the change (or difference) between these two supplementation conditions.
Change in muscle efficiency with beetroot juice supplementation | Day 8 (after 7 days of placebo supplementation) and day 29 (after 14 days of a washout period with no supplementation plus 7 days of beetroot juice supplementation)
  Muscle efficiency will be quantified as the ATP cost of contraction using phosphorus magnetic resonance spectroscopy (P-MRS). Muscle efficiency after 7 days of beetroot juice supplementation will be compared with muscle efficiency after 7 days of placebo supplementation, with the outcome measure being the change (or difference) between these two supplementation conditions.

OTHER OUTCOMES:
Change in plasma nitrate concentration with beetroot juice supplementation | Day 8 (after 7 days of placebo supplementation) and day 29 (after 14 days of a washout period with no supplementation plus 7 days of beetroot juice supplementation)
  Plasma nitrate concentration will be quantified using a nitrate colorimetric assay. Plasma nitrate concentration after 7 days of beetroot juice supplementation will be compared with plasma nitrate concentration after 7 days of placebo supplementation, with the outcome measure being the change (or difference) between these two supplementation conditions.
Change in plasma nitrite concentration with beetroot juice supplementation | Day 8 (after 7 days of placebo supplementation) and day 29 (after 14 days of a washout period with no supplementation plus 7 days of beetroot juice supplementation)
  Plasma nitrite concentration will be quantified using a nitrite colorimetric assay. Plasma nitrite concentration after 7 days of beetroot juice supplementation will be compared with plasma nitrite concentration after 7 days of placebo supplementation, with the outcome measure being the change (or difference) between these two supplementation conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No